CLINICAL TRIAL: NCT02891148
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 690517 in Healthy Male Subjects
Brief Title: Single Rising Dose Study of BI 690517 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1378.1; 2015-003642-10 (EudraCT Number)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy

ARMS (1):
- BI 690517 (Experimental)
  Interventions: Drug: BI 690517

INTERVENTIONS:
Drug: BI 690517
  Other Names: Vicadrostat

SUMMARY:
To investigate safety, tolerability, pharmacokinetics and pharmacodynamics following single rising doses of BI 690517

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and local legislation

Exclusion criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 60 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Values for serum sodium and potassium outside normal range at screening

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with adverse reactions, analysed as investigator defined drug-related adverse events. | From the first drug administration until end of the trial, up to 14 days
  The percentage of subjects with adverse reactions, analysed as investigator defined drug-related adverse events (AEs).

SECONDARY OUTCOMES:
Area under the concentration-time curve of the BI-690517 in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity) | Pharmacokinetic blood samples: 1:30 hours before drug administration and 30 minutes, 1, 1:30, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 hours after drug administration.
  Area under the concentration-time curve of the BI-690517 in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity).
Maximum measured concentration of the BI-690517 in plasma (Cmax) | PK blood samples: 1:30 hours before drug administration and 30 minutes, 1, 1:30, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 hours after drug administration.
  Maximum measured concentration of the BI-690517 in plasma (Cmax).

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany